CLINICAL TRIAL: NCT01682746
Title: Photodynamic Therapy (PDT) for Poor Prognosis Recurrent/Refractory Malignant Brain Tumors - A Phase I Study
Brief Title: Photodynamic Therapy (PDT) for Recurrent Pediatric Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Harry T Whelan, MD (Other)
Collaborators: Pinnacle Biologics Inc. (Industry)
Responsible Party: Sponsor-Investigator, Harry T Whelan, MD, Bleser Professor of Neurology, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 163588-1
Record Dates: First submitted 2012-09-05; First posted 2012-09-11 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Brain Tumor, Recurrent
Keywords: Brain Tumor; Photodynamic Therapy; Photochemotherapy; Astrocytoma; Pilocytic Astrocytoma; Low grade Astrocytoma; Anaplastic Astrocytoma; Glioblastoma; GBM; Chordoma; Germinoma; Germ Cell Tumor; Non-germinaoma; CNS Lymphoma; Craniopharyngioma; Brain Stem Glioma; Ependymoma; Mixed Glioma; Optic Nerve Glioma; Subependymoma; Medulloblastoma; Meningioma; Metastatic Brain Tumors; Oligodendroglioma; Pituitary Tumors; Primitive Neuroectodermal; PNET; Desmoplastic Neuroepithelial Tumor; DNET
MeSH Terms: conditions — Brain Neoplasms; Astrocytoma; Glioblastoma; Chordoma; Germinoma; Neoplasms, Germ Cell and Embryonal; Craniopharyngioma; Ependymoma; Glioma; Optic Nerve Glioma; Glioma, Subependymal; Medulloblastoma; Meningioma; Oligodendroglioma; Pituitary Neoplasms; Neuroectodermal Tumors, Primitive | interventions — Dihematoporphyrin Ether; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Photofrin (porfimer sodium) photodynamic therapy.
  Interventions: Drug: Photofrin (porfimer sodium) & photodynamic therapy.

INTERVENTIONS:
Drug: Photofrin (porfimer sodium) & photodynamic therapy. — Intravenous (IV) Photofrin
  This is a dose escalation study. Patients will receive Photofrin via an IV infusion approximately 24 hours prior to their tumor resection surgery and Photodynamic Therapy (PDT). Patients will be light sensitive immediately upon receiving the Photofrin and must observe photosensitivity & light precautions for a minimum of 30 days after the infusion.
  Photodynamic Therapy (PDT)
  After tumor resection, an optical fiber will be placed in the approximate center of the surgical cavity. Intralipid will be infused into the open tumor cavity while PDT is performed. The Intralipid will diffuse the light and ensure uniform delivery. Photoactivation of Photofrin is controlled by the total light dose delivered over the treatment time.

SUMMARY:
The goal of this proposal is to evaluate a new Photodynamic Therapy (PDT) modification which could revolutionize the treatment of brain tumors in children and adults. There are currently few cases published involving the use of PDT in infratentorial (in the posterior fossa) brain tumors in general and specifically those occurring in children. The investigators propose to test a technique, for the first time in the U.S., that demonstrated in Australian adult glioblastoma patients dramatic long-term, survival rates of 57% (anaplastic astrocytoma) and 37% (glioblastoma multiforme). These results are unprecedented in any other treatment protocol.

Photodynamic therapy (PDT) is a paradigm shift in the treatment of tumors from the traditional resection and systemic chemotherapy methods. The principle behind photodynamic therapy is light-mediated activation of a photosensitizer that is selectively accumulated in the target tissue, causing tumor cell destruction through singlet oxygen production. Therefore, the photosensitizer is considered to be the first critical element in PDT procedures, and the activation procedure is the second step. The methodology used in this proposal utilizes more intensive laser light and larger Photofrin photosensitizer doses than prior PDT protocols in the U.S. for brain tumor patients. The PDT will consist of photoillumination at 630 nm beginning at the center of the tumor resection cavity, and delivering a total energy of 240 J cm-2. The investigators feel that the light should penetrate far enough into the tissue to reach migrating tumor cells, and destroy these cells without harming the healthy cells in which they are dispersed.

The investigators will be testing the hypothesis that pediatric subjects with progressive/recurrent malignant brain tumors undergoing PDT with increased doses of Photofrin® and light energy than were used in our previous clinical study will show better progression free survival (PFS) and overall survival (OS) outcomes. PDT will also be effective against infratentorial tumors. The specific aims include determining the maximum tolerable dose (MTD) of Photofrin in children and looking for preliminary effectiveness trends.

ELIGIBILITY:
1. Age: ≥ 6 months and < 18 years
2. Disease: Patients with relapsed or refractory brain tumors are eligible. Patients must have had histologic verification of malignancy at original diagnosis or relapse. Tumors can be either supratentorial or infratentorial (posterior fossa) in location.
3. Disease Status: Patients must have potentially resectable disease.
4. Therapeutic Options: Patients' current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life.
5. Performance Level: Karnofsky 50% or greater for patients > 16 years of age and Lansky 50 or greater for patients < 16 years of age. Note: Neurologic deficits in patients with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
6. Predictable Life Expectancy: > 8 weeks
7. Prior Therapy: Patients must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy. At least 3 weeks from previous chemotherapy and 4 weeks from prior radiation therapy
8. Organ Function:

   Adequate bone marrow function

   Absolute neutrophil count ≥ 1,000

   Platelet count ≥ 100,000 (may transfuse to meet requirement)

   Adequate renal function

   Creatinine clearance or radioisotope GFR ≥ 70 mL/min/1.73 m2 OR

   A serum creatinine within normal range based on age/gender

   Adequate liver function Bilirubin (direct) ≤ 3X upper limit of normal (ULN) for age

   SGPT (ALT) ≤ 10X ULN

   For the purpose of this study, the ULN for SGPT is 45 U/L

   Serum albumin ≥ 2 g/dL

   Adequate coagulation

   PT and INR ≤ 2X ULN for age
9. Central Nervous System Function: Patients with seizure disorder may be enrolled if receiving non- enzyme inducing anticonvulsants and well controlled.
10. Informed Consent: All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.
11. Archival tumor tissue slides from initial diagnosis should be reviewed by CHW institutional pathologists prior to study enrollment whenever possible.

Exclusion Criteria

1. Disseminated disease (metastatic disease)
2. Pregnancy or Breast-Feeding: Pregnant or breast-feeding women will not be entered on this study, as risks of fetal and teratogenic adverse effects of Photofrin® are not known.
3. Other concurrent tumor therapy
4. Subjects with porphyria
5. Subjects taking potentially photosensitizing drugs
6. The presence of adverse events of neurologic function, photosensitivity, or photophobia Grade 4 or higher (CTCAE Version 4.0)
7. Allergy to eggs, soybean oil, or safflower oil (due to potential allergy against intralipids)
8. Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2013-03; Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Maximum tolerable dose (MTD) of Photofrin® in pediatric subjects | One to four weeks from PDT
  MTD is defined as the Photofrin® dose that precedes the dose level used with a subgroup of subjects that exhibits a greater than 33% DLT occurrence.
  DLT is defined as any of the following events with reasonable possibility to be attributable to the experimental intervention:
  1. Neurotoxicity: defined as a decline in neurological function manifest within 1 week of PDT and persistent to 4 weeks post-PDT. Adverse events of neurologic function of grade 4, or a level change from grade 1 to grade 3, within this period will constitute neurotoxicity for this study. The CTCAE V4.02 will be used.
  2. Photosensitivity: defined as a photosensitivity adverse event (CTCAE category dermatology/skin) of grade 4 occurring within the same period.
  3. Ocular sensitivity: Photofrin®-induced ocular sensitivity is defined as a photophobia adverse event (CTCAE category ocular/visual) of grade 4 within the same period.
  4. Any other toxicity of CTCAE grade 4 or higher within the same period.

SECONDARY OUTCOMES:
Brain tumor response | Response ocurring within 3 years after PDT
  To preliminarily define the antitumor activity of Photofrin and laser light activation within the confines of a Phase 1 Study. We will follow progression free survival and overall survival for 3 years post PDT treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Harry T Whelan, MD, Principal Investigator — Medical College of Wisconsin; Jeff Knipstein, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Wauwatosa, Wisconsin, United States